CLINICAL TRIAL: NCT00187252
Title: Management of Atrial Fibrillation Suppression in AF-HF COmorbidity Therapy
Brief Title: Mascot Study: Management of Atrial Fibrillation (AF) Suppression in AF-Heart Failure (HF) COmorbidity Therapy
Acronym: MASCOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Christophe Bailleul, St. Jude Medical
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR03001HF
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; Atrial Fibrillation; Ventricular Dysfunction
Keywords: Ventricular Dyssynchrony
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation; Ventricular Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CRT + AF Suppression turned ON
  Interventions: Device: Atrial Overdrive Pacing
- 2 (Active Comparator): CRT + AF Suppression turned OFF
  Interventions: Device: Atrial Overdrive Pacing

INTERVENTIONS:
Device: Atrial Overdrive Pacing — Pacemaker/ ICD implant

SUMMARY:
The purpose of this study is to evaluate whether adding AF Suppression™ to cardiac resynchronization therapy (CRT) improves the prognosis of heart failure patients benefiting from cardiac resynchronization therapy.

ELIGIBILITY:
Inclusion Criteria:

* HF patients
* New York Heart Association (NYHA) III - IV
* Spontaneous QRS ≥130 ms and/or mechanical interventricular delay > 50 ms
* Left ventricular ejection fraction (LVEF) ≤ 35%
* Left ventricular end diastolic diameter (LVEDD) ≥ 55 mm
* Optimized medical regimen
* Age > 18 years

Exclusion Criteria:

* Unstable angina or acute myocardial infarction (MI) (< 3 months)
* Coronary artery bypass grafting (CABG) or percutaneous transluminal coronary angioplasty (PTCA) < 3 months
* Life expectancy < 6 months

  * Permanent AF
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2003-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of permanent atrial fibrillation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Padeletti, MD, Principal Investigator — Ospedale Carregi, Firenze, Italy
Locations (1):
- Clinica Medica Generale e Cardiologia - Ospedale Careggi, Florence, Italy

REFERENCES:
- [Background] Padeletti L, Musilli N, Porciani MC, Colella A, Di Biase L, Ricciardi G, Pieragnoli P, Michelucci A, Gensini G. Atrial fibrillation and cardiac resynchronization therapy: the MASCOT study. Europace. 2004 Sep;5 Suppl 1:S49-54. doi: 10.1016/j.eupc.2004.07.007. PMID 15450280
- [Derived] Padeletti L, Muto C, Maounis T, Schuchert A, Bongiorni MG, Frank R, Vesterlund T, Brachmann J, Vicentini A, Jauvert G, Tadeo G, Gras D, Lisi F, Dello Russo A, Rey JL, Boulogne E, Ricciardi G; Management of Atrial fibrillation Suppression in AF-HF COmorbidity Therapy Study Group. Atrial fibrillation in recipients of cardiac resynchronization therapy device: 1-year results of the randomized MASCOT trial. Am Heart J. 2008 Sep;156(3):520-6. doi: 10.1016/j.ahj.2008.04.013. Epub 2008 Jul 7. PMID 18760135